CLINICAL TRIAL: NCT03360175
Title: Correlation of Eicosanoid and Proresolving Lipid Mediator Temporal Profiles and Resolution of Pain After Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mieke A. Soens, MD Staff Anesthesiologist, Brigham and Women's Hospital
Other Study IDs: 2017P002402
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained for determination of pro-inflammatory/ pro resolving lipid mediator temporal profiles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic Surgery Patients: Inclusion criteria include: Patients scheduled to undergo thoracic surgery at Brigham and Women's Hospital, between the ages 18-85 years old. Exclusion criteria are: pre-existing chronic pain or opioid use; current treatment with corticosteroids; evidence of active infection; chronic liver disease; end-stage renal disease (CKD-5); chronic inflammatory disorders; recent major surgery or illness within 30 days; use of immunosuppressive medication; history of organ transplantation.
  Pro-inflammatory eicosanoid and pro resolving lipid mediator temporal profiles will be determined pre-operatively, on post-operative day 1 and on post-operative day 14. In addition, daily pain scores will be recorded for 60 days after surgery and at 3, 6 and 12 months.
  Interventions: Other: No intervention - observational study

INTERVENTIONS:
Other: No intervention - observational study — No intervention - observational study

SUMMARY:
The aim of the current pilot study is to investigate whether perioperative dysregulated systemic lipid mediator pathways (more specifically increased pro-inflammatory and decreased anti-inflammatory pathways) are associated with slower resolution of pain after surgery and increased risk for development of persistent postsurgical pain (PPSP). In addition, we will look for correlations between the pro-resolving lipid mediator profile and Quality of Recovery (QoR-15), duration of hospital stay, and frequency of complications, e.g. wound infections.

DETAILED DESCRIPTION:
This is a prospective, observational pilot study that will assess whether 1) a peri-operative dysregulated metabolo-lipidomics or SPM profile is associated with slower resolution of pain after surgery and an increased risk for development of persistent postsurgical pain (PPSP), and 2) whether a peri-operative dysregulated metabolo-lipidomics profile correlates with low Quality of Recovery (QoR-15) scores, duration of hospital stay and frequency of complications, e.g. wound infection.

The study will address the following Specific Aims:

Specific Aim 1: To determine the correlation between the perioperative eicosanoid and pro-resolving lipid mediator temporal profile and day-to-day resolution of pain after thoracic surgery.

We hypothesize that patients who have slower resolution of pain after thoracic surgery have dysregulated systemic lipid mediator pathways when compared to those patients who have faster resolution of pain.

Specific Aim 2: To determine the effectiveness of perioperative SPM signature as a novel predictive marker for the development of persistent pain after surgery (PPSP).

We hypothesize that patients with dysregulated systemic lipid mediator pathways, more specifically up-regulated pro-inflammatory lipid mediator pathways and down-regulated pro-resolving lipid mediator pathways, are more likely to develop PPSP.

Specific Aim 3: To determine the correlation between the perioperative eicosanoid and pro-resolving lipid mediator temporal profile and quality of recovery after surgery, duration of hospital stay and complications.

We hypothesize that dysregulated lipid mediator profiles are associated with a decreased Quality of Recovery Score (QoR-15), prolonged hospital stay and increased rates of complications, such as problems with wound healing and infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Patients scheduled to undergo thoracic surgery at Brigham and Women's Hospital

Exclusion Criteria:

* Pre-existing chronic pain or opioid use
* Current treatment with corticosteroids
* Evidence of active infection
* Chronic liver disease, end-stage renal disease (CKD-5), or chronic inflammatory disorders
* Recent major surgery or illness within 30 days
* Use of immunosuppressive medication
* History of organ transplantation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo thoracic surgery at Brigham and Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-12-11 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
time course of pain resolution after thoracic surgery | 12 months

SECONDARY OUTCOMES:
incidence of persistent pain after thoracic surgery | 18 months
Quality of Recovery after thoracic surgery | 12 months

IPD SHARING:
Plan to Share IPD: No